CLINICAL TRIAL: NCT02888678
Title: A Randomized Study Evaluating an Intervention Integrating Economic Strengthening and HIV Prevention Programs for Vulnerable Youth in South Africa
Brief Title: Evaluation of an Integrated Economic Strengthening and HIV Prevention Program for Vulnerable Youth in South Africa
Acronym: ASPIRES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Foundation for Professional Development (Unknown); Future Families (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 741818
Record Dates: First submitted 2016-06-17; First posted 2016-09-05 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: HIV; HIV Infections
Keywords: ASPIRES
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ES + HIV Prevention (Experimental): Economic Strengthening + HIV prevention education combined intervention consists of 2 parts.
  Impumelelo: This intervention consists of 15 one-hour long sessions on financial education in combination with access to appropriate youth-friendly savings mechanisms.
  Vhutshilo 2.2: . This intervention consists of 15 one-hour long sessions that are interactive, skills focused, and cover such topics as expressing one's feelings; dealing with loss and grief; decision-making; coping; gender violence; understanding HIV and other sexually transmitted infections; healthy relationships and staying safe in sexual relationships; and contraception and risks associated with unplanned pregnancy.
  Interventions: Behavioral: Economic Strengthening (Impumelelo); Behavioral: HIV Prevention Education (Vhutshilo 2.2)
- ES only (Experimental): Economic Strengthening (Impumelelo): This intervention consists of 15 one-hour long sessions on financial education in combination with access to appropriate youth-friendly savings mechanisms.
  Interventions: Behavioral: Economic Strengthening (Impumelelo)
- HIV only (Experimental): HIV Prevention Education (Vhutshilo 2.2): This intervention consists of 15 one-hour long sessions that are interactive, skills focused, and cover such topics as expressing one's feelings; dealing with loss and grief; decision-making; coping; gender violence; understanding HIV and other sexually transmitted infections; healthy relationships and staying safe in sexual relationships; and contraception and risks associated with unplanned pregnancy.
  Interventions: Behavioral: HIV Prevention Education (Vhutshilo 2.2)
- No intervention (control) (No Intervention): The control group will not receive the ES or HIV prevention interventions. They will receive the basic package of services available to all beneficiaries of Future Families.

INTERVENTIONS:
Behavioral: Economic Strengthening (Impumelelo) — Economic Strengthening (Impumelelo): This intervention consists of 15 one-hour long sessions on financial education in combination with access to appropriate youth-friendly savings mechanisms.
  Arms: ES + HIV Prevention; ES only
Behavioral: HIV Prevention Education (Vhutshilo 2.2) — HIV Prevention Education (Vhutshilo 2.2): This intervention consists of 15 one-hour long sessions that are interactive, skills focused, and cover such topics as expressing one's feelings; dealing with loss and grief; decision-making; coping; gender violence; understanding HIV and other sexually transmitted infections; healthy relationships and staying safe in sexual relationships; and contraception and risks associated with unplanned pregnancy.
  Arms: ES + HIV Prevention; HIV only

SUMMARY:
This study evaluates whether the integration of an Economic Strengthening program with an HIV-prevention education program produce synergistic effects on economic and health outcomes for South African youth ages 14-17 years old.

DETAILED DESCRIPTION:
In South Africa, the overall HIV prevalence of 12.2% can be reviewed based on a number of factors: age, province, type of locality, race, economic household conditions, and marital status. Those to be reached through the ASPIRES intervention and evaluation are economically disadvantaged Black African youth, male and female, located in urban localities in Gauteng province, and are situated within a setting of high risk and vulnerability for HIV. The ASPIRES project is providing technical assistance to provide economic strengthening (ES) and HIV prevention education programming for adolescents. The ASPIRES ES intervention includes financial capability building through the provision of financial education in combination with access to appropriate youth-friendly savings mechanisms. The HIV prevention education intervention Vhutshilo 2.2 will be used in this study.

This study will assess whether the integration of an ES intervention with an HIV-prevention education intervention improves economic and health outcomes beyond singular interventions, estimate the resources required at the program level to support the ES and HIV-prevention education interventions; and describe whether the interventions were perceived as effective in addressing economic and health outcomes and to describe how and why the interventions were perceived as effective or not.

This study will enroll up to 2000 youth ages 14-17 and randomly assign them to either 1) ES intervention only, 2) HIV prevention intervention only, 3) combined ES and HIV intervention, or 4) no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Beneficiary of Future Families in a study community
* Parent or guardian consent allowing adolescent to participate in the study
* Willing to sign or make their mark on an assent form
* Willing to provide contact information
* Only one adolescent is eligible per household

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1773 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
STI prevalence Endline 1 | Nine months after baseline interview
  Prevalence of gonorrhea, trichomoniasis or chlamydia infection (lab report)
STI prevalence Endline 2 | eighteen months after baseline interview
  Prevalence of gonorrhea, trichomoniasis or chlamydia infection (lab report)

SECONDARY OUTCOMES:
Prevalence of pregnancy Endline 1 | Nine months after baseline interview
  Prevalence of pregnancy among female participants (lab report)
Prevalence of pregnancy Endline 2 | eighteen months after baseline interview
  Prevalence of pregnancy among female participants (lab report)
Percent of adolescents engaging in protective sexual behavior Endline 1 | In the 6 month time period prior to the date of the follow up visit
  Percent of adolescents engaging in protective sexual behavior, defined as self-reported abstinence or consistent condom use (a condom used every time) over the past 6 months
Percent of adolescents engaging in protective sexual behavior Endline 2 | In the 6 month time period prior to the date of the follow up visit
  Percent of adolescents engaging in protective sexual behavior, defined as self-reported abstinence or consistent condom use (a condom used every time) over the past 6 months
Percent of adolescents engaging in transactional sex in past 6 months Endline 1 | In the 6 months prior to the date of the follow up visit
  self-reported
Percent of adolescents engaging in transactional sex in past 6 months Endline 2 | In the 6 months prior to the date of the follow up visit
  self-reported
Percent of adolescents reporting two or more sexual partners in the past 6 months Endline 1 | In the 6 months prior to the date of the follow up visit
  self-reported
Percent of adolescents reporting two or more sexual partners in the past 6 months Endline 2 | In the 6 months prior to the date of the follow up visit
  self-reported
Mean HIV knowledge score Endline 1 | Nine months after baseline interview
  HIV knowledge score calculated based on the answers to survey questions
Mean HIV knowledge score Endline 2 | Eighteen months after baseline interview
  HIV knowledge score calculated based on the answers to survey questions
Mean financial literacy score Endline 1 | Nine months after baseline interview
  Financial literacy score calculated based on the answers to survey questions
Mean financial literacy score Endline 2 | eighteen months after baseline interview
  Financial literacy score calculated based on the answers to survey questions
Percent of adolescents participating in savings group Endline 1 | Nine months after baseline interview
  Percent of adolescents participating in savings group (self report)
Percent of adolescents participating in savings group Endline 2 | eighteen months after baseline interview
  Percent of adolescents participating in savings group (self report)
Percent of adolescents opening savings account Endline 1 | Nine months after baseline interview
  Percent of adolescents opening savings account (self report)
Percent of adolescents opening savings account Endline 2 | eighteen months after baseline interview
  Percent of adolescents opening savings account (self report)
Mean total amount of savings in past 1 year Endline 1 | In the one year prior to the date of the 9 month follow up visit
  Mean total amount of savings starting from prior to enrollment in the study up to 9 months of participation in the study
Mean total amount of savings in past 1 year Endline 2 | In the one year prior to the date of the 18 month follow up visit
  Mean total amount of savings in past 1 year reported by adolescents (self report)
Percent of adolescents saving for education Endline 1 | Nine months after baseline interview
  Percent of adolescents saving for education (self report)
Percent of adolescents saving for education Endline 2 | eighteen months after baseline interview
  Percent of adolescents saving for education (self report)
Percent of adolescents whose caregiver provided money for savings Endline 1 | Nine months after baseline interview
  Percent of adolescents whose caregiver provided money for savings (self report)
Percent of adolescents whose caregiver provided money for savings Endline 2 | eighteen months after baseline interview
  Percent of adolescents whose caregiver provided money for savings (self report)
Percent of adolescents who participate in household budgeting Endline 1 | Nine months after baseline interview
  Percent of adolescents who participate in household budgeting (self report)
Percent of adolescents who participate in household budgeting Endline 2 | eighteen months after baseline interview
  Percent of adolescents who participate in household budgeting (self report)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Burke, PhD, Principal Investigator — FHI 360
Locations (1):
- community Based Recruitment, Pretoria, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burke HM, Chen M, Murray K, Bezuidenhout C, Ngwepe P, Bernholc A, Medina-Marino A. The effects of the integration of an economic strengthening and HIV prevention education programme on the prevalence of sexually transmitted infections and savings behaviours among adolescents: a full-factorial randomised controlled trial in South Africa. BMJ Glob Health. 2020 Apr 7;5(4):e002029. doi: 10.1136/bmjgh-2019-002029. eCollection 2020. PMID 32355569